CLINICAL TRIAL: NCT04158622
Title: A Randomized controllEd Trial Comparing Pneumatic Retinopexy Versus Pars plAna Vitrectomy for the Management of Primary Retinal Detachment: Retinal Displacement Rates and Impact on Patient Quality of Life: The REVEAL Study
Brief Title: Retinal Displacement Rates in Pneumatic Retinopexy Versus Pars Plana Vitrectomy For Primary Retinal Detachment
Acronym: REVEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-239
Record Dates: First submitted 2019-10-16; First posted 2019-11-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Retinal Detachment; Metamorphopsia
MeSH Terms: conditions — Retinal Detachment; Vision Disorders | interventions — Lasers; Cryotherapy; Predictive Value of Tests

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumatic Retinopexy (Experimental): Patients with retinal detachment allocated to pneumatic retinopexy + laser/cryotherapy
  Interventions: Procedure: PnR + laser/cryotherapy
- Pars Plana Vitrectomy (Experimental): Patients with retinal detachment allocated to pars plana vitrectomy + laser/cryotherapy
  Interventions: Procedure: PPV + laser/cryotherapy

INTERVENTIONS:
Procedure: PnR + laser/cryotherapy — Pneumatic retinopexy plus laser/cryotherapy
  Arms: Pneumatic Retinopexy
Procedure: PPV + laser/cryotherapy — Pars plana vitrectomy plus laser/cryotherapy
  Arms: Pars Plana Vitrectomy

SUMMARY:
Patients may experience metamorphopsia, or image distortion, after having vitrectomy to repair their rhegmatogenous retinal detachments (RRDs) especially those with a detached macula. Retinal displacement, as measured on autofluorescence photography, likely contributes to this distortion. There is no study in the scientific literature comparing the rate of retinal displacement and its association with visual function, including metamorphopsia, in patients undergoing different procedures for RRD repair. Based on the recently published PIVOT trial, patients who underwent Pneumatic Retinopexy (PnR) had less vertical distortion at 12 months than patients who had Pars Plana Vitrectomy (PPV). It is hypothesized that PnR will cause less retinal displacement than PPV for patients with macula-off primary retinal detachment.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachments (RRD) are a sight-threatening condition with an incidence of approximately 10 per 100 000 people. RRDs can be broadly classified into those with the macula still attached, and those with the macula detached. Without surgical intervention by a vitreoretinal surgeon, retinal detachment almost invariably results in permanent sight loss. Current techniques for RRD repair include scleral buckle (SB), pneumatic retinopexy (PnR), and pars plana vitrectomy (PPV) with or without combination of SB.

Pneumatic retinopexy (PnR) is a minor surgical intervention employed to repair retinal detachments, carried out in the clinic's procedure room. Standard criteria for this procedure include one or more retinal breaks within one clock hour located at the superior eight clock hours, without signs of proliferative vitreoretinopathy. The procedure involves injection of a small gas bubble into the eyeball via a fine needle. Two gases can be injected into the eye: perfluoropropane (C3F8), which lasts 6 weeks, and sulfur hexafluoride (SF6), which lasts about 2 weeks. After injection of the gas bubble, the patient is required to maintain a strict 'head posture' (for example, head tilt to left) for up to 10 days. The gas bubble spontaneously dissipates after 2-6 weeks, depending on the gas selected. Additionally, laser treatment or cryotherapy is carried out either before or 1-2 days after injection of the gas bubble, to secure the retinal tear. The advantages of PnR over PPV are: (1) Low risk of cataract - secondary cataract formation is uncommon after PnR, but more common after PPV; (2) Quicker visual rehabilitation - due to the smaller size gas bubble and less invasive nature of the procedure, patients undergoing PnR commonly have improved vision within days after treatment; (3) Immediate availability of intervention - unlike PPV, PnR is carried out in a treatment room, and there are no delays due to operating room availability.

Pars plana vitrectomy (PPV) is a surgical procedure carried out in the operating room under regional anesthetic, and often times sedation. During PPV, the vitreous gel is removed from the eye to allow space for a larger gas bubble than is possible in PnR, and also to relieve any vitreous traction which may otherwise impair reattachment of the retina. The retina is reattached by either draining the subretinal fluid through a peripheral retinal break; by draining the subretinal fluid through a posterior retinotomy; or by using a heavier-than-water liquid such as perfluocarbon (PFC) to push out the subretinal fluid. Laser or cryotherapy is applied around the retinal tear to create chorioretinal adhesions (as in PnR). At the end of the surgery, the vitreous cavity is filled with a substance that will tamponade the retina to the wall of the eye while the adhesions form. Tamponade agents can be temporary, such as SF6 and C3F8 (same gases as mentioned for PnR), which are absorbed by 2-6 weeks, or long term, such as silicone oil, which requires a second surgery to remove. After the surgery, the patient may be required to maintain a 'head posture' (for example, head tilt to left) for up to one week to support the area of the retinal tear optimally by 'floating' the gas bubble up against it. As the gas bubble is larger in PPV, the head posturing requirements are less strict. The advantages of PPV over PnR are: (1) higher primary single procedure success rate (although same final reattachment success rate); (2) less follow-up visits in the first week.

Patients may experience metamorphopsia, or image distortion, after having their RRD repaired especially those with a detached macula. In 2010, Shiragami et al were the first to demonstrate hyperfluorescent lines, adjacent to the retinal blood vessels in Fundus autofluorescence imaging (FAF) of the retina after RD repair surgery.They theorized that these lines which are called Retinal Vessel Printings (RVP) correspond to the location of the retinal blood vessels before the retinal detachment. In FAF, an image is taken with structures that naturally fluoresce such as the lipofuscin in the retinal pigment epithelium (RPE) appearing brighter. According to this theory, prior to the retinal detachment, certain RPE cells were covered by the retinal blood vessels. Afterwards, with the displacement of the retina due to the retinal detachment these RPE cells become exposed to light which increases in metabolic activity producing more lipofuscin and therefore, appearing more hyperautofluorescent on the FAF. Moreover, these reference lines allow us to quantify the displacement of the retina after retinal detachment surgeries. In this study by Shiragami, 62.8% of eyes demonstrated hyperautofluorescent lines superior to the retinal blood vessels suggesting downward displacement. Since Shiragami's first report, several other studies looked into retinal displacement after RD repair.

There is no study in the scientific literature comparing the rate of retinal displacement and its association with visual function, including metamorphopsia, in patients undergoing different procedures for RRD repair.

The aim of this study is to compare retinal displacement following primary macula-off retinal detachment repair treated with pneumatic retinopexy (PnR) versus pars plana vitrectomy (PPV). The primary study hypothesis is that pneumatic retinopexy will cause less retinal displacement at 3 months for patients with macula-off primary retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Macula-off retinal detachment
* Single retinal break OR group of breaks no larger than four clock hours apart between each other (Figure 2)
* All breaks in detached retina must be between 3-9 o'clock (Figure 2, blue lines)
* No significant proliferative vitreoretinopathy (PVR) (can have grade A or B)

Exclusion Criteria:

* Inferior breaks in detached retina. NOTE: Patient can have any number, location and size of retinal breaks or lattice degeneration in attached retina.
* Inability to read English language
* Age < 18 years
* Mental incapacity
* Previous vitrectomy (index eye)
* Previous retinal detachment (index eye)
* Previous or concurrent retina pathology (e.g. vascular)
* Previous or concurrent macula pathology (macular hole, ERM, AMD, DME)
* Anterior segment surgery within 3 months
* Inability to maintain post intervention head positioning
* Inability to carry out detailed examination of the peripheral retina due to media opacity NOTE: Lens/posterior hyaloid status does not impact eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Retinal Displacement | 3 months post intervention
  Retinal displacement by the presence of retinal vessels printing on FAF imaging

SECONDARY OUTCOMES:
Visual acuity (ETDRS) | 3, 6, and 12 months post intervention
  The Early Treatment of Diabetic Retinopathy Study (ETDRS) developed a vision chart that has now become the gold standard for measuring visual function in ophthalmic research.
Objective Metamorphopsia | 3, 6, and 12 months post intervention
  Metamorphopsia assessed by M-CHARTS, which measures the minimum visual angle of a dotted line needed to detect metamorphopsia.
Subjective Metamorphopsia | 3, 6, and 12 months post intervention
  Metamorphopsia Questionnaire; The Questionnaire is a valid tool to assess patient's subjective perception of metamorphopsia. The minimum score is 0 and maximum score is 3, and higher scores mean a worse outcome.
Aniseikonia Test | 3, 6, and 12 months post intervention
  Aniseikonia Test measures the ratio of image size difference between the 2 eyes.
Optical Coherence Tomography (OCT) cystoid macular edema (CME) | 3, 6, and 12 months post intervention
  Two readers will analyze the cross-sectional OCT images regarding the presence of CME.
Optical Coherence Tomography (OCT) layers disruption | 3, 6, and 12 months post intervention
  Two readers will analyze the cross-sectional OCT images regarding the presence of retinal layers disruption.
Optical Coherence Tomography (OCT) retinal folds | 3, 6, and 12 months post intervention
  Two readers will analyze the cross-sectional OCT images regarding the presence of outer/inner retinal folds.
Optical Coherence Tomography Angiography (OCTA) capillary perfusion | 3, 6, and 12 months post intervention
  Two readers will analyze OCTA images regarding retinal capillary plexuses perfusion.
Optical Coherence Tomography Angiography (OCTA) changes | 3, 6, and 12 months post intervention
  Two readers will analyze OCTA images regarding area of foveal avascular zone.
Association between retinal displacement (RVP) and visual function (ETDRS) | 3 months post intervention
  Association between the presence of retinal displacement and ETDRS values.

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, FRSCS, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Eye Clinic, Toronto, Ontario, Canada